CLINICAL TRIAL: NCT01634789
Title: A Phase 1, Open-label, Single-dose, Randomized, 4-treatment, 4- Period, Crossover, Pilot Bioavailability Study of 3 Test Tablet Formulations of Bazedoxifene (Bza) Compared With A Reference Tablet Formulation of Bza/Conjugated Estrogens (ce) in Healthy Postmenopausal Women
Brief Title: A Pilot Bioavailability Study of 3 Test Tablet Formulations of Bazedoxifene Compared With A Reference Tablet Formulation of Bazedoxifene/Conjugated Estrogens in Healthy Postmenopausal Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated on 10 December 2012 due to low enrollment. The decision to terminate the study was not based on safety or efficacy issues.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2311014; 3115B1-1146
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: bioavailability
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test Treatment 1: bazedoxifene (Experimental): Test Treatment 1
  Interventions: Drug: bazedoxifene
- Test Treatment 2: bazedoxifene (Experimental): Test Treatment 2
  Interventions: Drug: bazedoxifene
- Test Treatment 3: bazedoxifene (Experimental): Test Treatment 3
  Interventions: Drug: bazedoxifene
- Reference Treatment: bazedoxifene/conjugated estrogens (Experimental): Reference Treatment
  Interventions: Drug: bazedoxifene/conjugated estrogens

INTERVENTIONS:
Drug: bazedoxifene — 20 mg oral tablet, single dose
  Other Names: TSE-424
  Arms: Test Treatment 1: bazedoxifene
Drug: bazedoxifene — 20 mg oral tablet, single dose
  Other Names: TSE-424
  Arms: Test Treatment 2: bazedoxifene
Drug: bazedoxifene — 20 mg oral tablet, single dose
  Other Names: TSE-424
  Arms: Test Treatment 3: bazedoxifene
Drug: bazedoxifene/conjugated estrogens — 20 mg / 0.625 mg oral tablet, single dose
  Other Names: BZA/CE
  Arms: Reference Treatment: bazedoxifene/conjugated estrogens

SUMMARY:
The purpose of this study is to evaluate 3 test formulations relative to a reference formulation.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy postmenopausal women
* Body mass index (BMI) in the range of 18.0 to 35.0 kg/m2 and body weight >= 50 kg

Exclusion Criteria:

* Pregnant or nursing females; females of childbearing potential

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose
Area Under the Concentration-Time Curve from Time 0 to Last Observable Concentration (AUCT) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose
Time of Maximum Plasma Concentration (Tmax) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose
Elimination-phase Half-life (t1/2) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose
Relative Bioavailability (F) | 0, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 9, 16, 24, 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2311014&StudyName=A%20Pilot%20Bioavailability%20Study%20of%203%20Test%20Tablet%20Formulations%20of%20Bazedoxifene%20Compared%20with%20A%20Reference%20Tablet%20Formulation%20of%20Bazedoxifene/C